CLINICAL TRIAL: NCT01282424
Title: A Phase 2 Study to Assess the Efficacy and Safety of Idelalisib in Subjects With Indolent B-Cell Non-Hodgkin Lymphomas Refractory to Rituximab and Alkylating Agents
Brief Title: Efficacy and Safety Study of Idelalisib in Participants With Indolent B-Cell Non-Hodgkin Lymphomas
Acronym: DELTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-09; 2010-022155-33 (EudraCT Number)
Record Dates: First submitted 2011-01-21; First posted 2011-01-25 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-06

CONDITIONS: Follicular Lymphoma; Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma; Marginal Zone Lymphoma
Keywords: indolent Non-Hodgkin Lymphoma; Non-Hodgkin Lymphoma; iNHL; NHL; GS-1101; CAL-101; PI3K; Phosphatidylinositol 3-kinase; Follicular Lymphoma (FL); Small lymphocytic lymphoma (SLL); Lymphoplasmacytoid lymphoma (LPL); Marginal zone lymphoma (MZL)
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin; Waldenstrom Macroglobulinemia | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idelalisib (Experimental): Treatment with idelalisib will be continued until tumor progression or development of unacceptable toxicity.
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib 150 mg tablet administered orally twice daily
  Other Names: Zydelig®; GS-1101; CAL-101; IDELA

SUMMARY:
The primary objective will be to assess the overall response rate and to evaluate the efficacy and safety of idelalisib (IDELA; GS-1101) in participants with previously treated indolent Non-Hodgkin Lymphoma (iNHL) that is refractory both to rituximab and to alkylating-agent-containing chemotherapy.

Eligible participants will initiate oral therapy with idelalisib at a starting dose of 150 mg taken twice per day. Treatment with idelalisib can continue in compliant participants as long as the study is still ongoing and the participants appear to be benefiting from treatment with acceptable safety.

ELIGIBILITY:
Key Inclusion Criteria:

* Karnofsky performance status of ≥ 60 (Eastern Cooperative Oncology Group [ECOG] performance score of 0, 1, or 2)
* Histologically confirmed diagnosis of B-cell iNHL, with histological subtype limited to the following:

  * Follicular lymphoma (FL)
  * Small lymphocytic lymphoma (SLL) with absolute lymphocyte count < 5 x 10^9/L at the time of diagnosis and on baseline laboratory assessment performed within 4 weeks prior to the start of study drug administration
  * Lymphoplasmacytic lymphoma (LPL), with or without associated Waldenstroms Macroglobulinemia (WM)
  * Marginal zone lymphoma (MZL) (splenic, nodal, or extranodal)
* Prior treatment with ≥ 2 prior chemotherapy-based or immunotherapy-based regimens for iNHL
* Presence of radiographically measurable lymphadenopathy or extranodal lymphoid malignancy
* Prior treatment with rituximab and with an alkylating agent (eg, bendamustine, cyclophosphamide, ifosfamide, chlorambucil, melphalan, busulfan, nitrosoureas) for iNHL
* Lymphoma that is refractory to rituximab and to an alkylating agent
* Discontinuation of all other therapies for treatment of iNHL ≥ 3 weeks before Visit 2
* For men and women of childbearing potential, willingness to abstain from sexual intercourse or employ an effective method of contraception during the study drug administration and follow-up periods
* Willingness and ability to provide written informed consent and to comply with the protocol requirements

Key Exclusion Criteria:

* Central nervous system or leptomeningeal lymphoma
* Known histological transformation from iNHL to diffuse large B-cell lymphoma
* History of a non-lymphoma malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, localized prostate cancer, other adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for ≥ 5 years
* Evidence of ongoing systemic bacterial, fungal, or viral infection (excluding viral upper respiratory tract infections) at the time of initiation of study treatment
* Pregnancy or breastfeeding
* Ongoing alcohol or drug addiction
* Known history of drug-induced liver injury, chronic active hepatitis B infection, chronic active hepatitis C infection, alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by stones, cirrhosis of the liver, or portal hypertension
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy, including systemic corticosteroids. Participant may be using topical or inhaled corticosteroids.
* Prior therapy with idelalisib
* Exposure to another investigational drug within 3 weeks prior to start of study treatment
* Concurrent participation in another therapeutic treatment trial
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, ECG finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the participant, alter the absorption, distribution, metabolism or excretion of the study drug, or impair the assessment of study results

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-03-18 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (41):
- United States (22):
  - St. Jude Medical Center, Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA, Los Angeles, California
  - Central Coast Medical Oncology, Santa Maria, California
  - Stanford Cancer Center, Stanford, California
  - Collaborative Research Group, LLC, Boynton Beach, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center Hackensack University Medical Center, Hackensack, New Jersey
  - University of Medicine and Dentistry of NJ, New Brunswick, New Jersey
  - Weill Cornell -New York Presbyterian Hospital, New York, New York
  - Montefiore Medical Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Chattanooga Hem/Oncology Ass (SCRI), Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- France (4):
  - CHU Morvan, Brest
  - Centre Hospitalier de Lyon Sud, Pierre-Bénite
  - Centre Henri Bequerel, Rouen
  - CHU Bretonneau - Centre Kaplan, Tours
- Germany (4):
  - Charité Campus Virchow Klinikum, Berlin
  - Universitätsklinikum Essen, Essen
  - Klinikum der Universität München-Großhadern, München
  - Universitatsklinikum Ulm, Ulm
- Italy (4):
  - Azienda Ospedaliera di Bologna - Policlinico S. Orsola Malpighi, Bologna
  - A.O.U. San Martino, Genova
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Università "Sapienza", Rome
- Poland (2):
  - Małopolskie Centrum Medyczne, Krakow
  - Centrum Onkologii w Warszawie, Warsaw
- United Kingdom (5):
  - St James's Institute of Oncology, Leeds
  - St Bartholemews Hospital, London
  - Sarah Cannon Institute, London
  - The Christie Hospital, Manchester
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Result] Salles GA, Kahl, BS, Wagner-Johnston ND, et al. Interim results from a phase 2 study of PI3Kδ inhibitor idelalisib in patients with relapsed indolent non-Hodgki lymphoma (iNHL) refractory to both rituximab and an alkylating agent. 12th International Conference on Malignant Lymphoma, Palazzo dei Congressi, Lugano, Switzerland, June 19-22, 2013 Abstract No: 064bis.
- [Result] Gopal AK, Kahl BS, de Vos S, Wagner-Johnston ND, Schuster SJ, Jurczak WJ, Flinn IW, Flowers CR, Martin P, Viardot A, Blum KA, Goy AH, Davies AJ, Zinzani PL, Dreyling M, Johnson D, Miller LL, Holes L, Li D, Dansey RD, Godfrey WR, Salles GA. PI3Kdelta inhibition by idelalisib in patients with relapsed indolent lymphoma. N Engl J Med. 2014 Mar 13;370(11):1008-18. doi: 10.1056/NEJMoa1314583. Epub 2014 Jan 22. PMID 24450858
- [Derived] Ma S, Chan RJ, Gu L, Xing G, Rajakumaraswamy N, Ruzicka BB, Wagner-Johnston ND. Retrospective Analysis of the Impact of Adverse Event-Triggered Idelalisib Interruption and Dose Reduction on Clinical Outcomes in Patients With Relapsed/Refractory B-Cell Malignancies. Clin Lymphoma Myeloma Leuk. 2021 May;21(5):e432-e448. doi: 10.1016/j.clml.2020.12.016. Epub 2020 Dec 24. PMID 33516721
- [Derived] Barrientos JC, Hillmen P, Salles G, Sharman J, Stilgenbauer S, Gurtovaya O, Xing G, Ruzicka B, Bhargava P, Ghia P, Pagel JM. No increased bleeding events in patients with relapsed chronic lymphocytic leukemia and indolent non-Hodgkin lymphoma treated with idelalisib. Leuk Lymphoma. 2021 Apr;62(4):837-845. doi: 10.1080/10428194.2020.1845339. Epub 2020 Dec 10. PMID 33297794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 54 study sites in North America and Europe. The first participant was screened on 04 March 2011. The last participant observation was on 16 May 2018.
Pre-assignment Details: 125 participants were enrolled and treated and comprise the Intent-to-Treat (ITT) Analysis Set.
Groups:
- Idelalisib: Idelalisib 150 mg tablet administered orally twice daily until tumor progression or development of unacceptable toxicity.
Period: Treatment Period (TP) (81 Months)
Arm/Group | Idelalisib
Started | 125
Completed: Disease Progression | 70
Completed: Death | 9
Completed | 79
Not Completed | 46
Not completed — Adverse Event | 30
Not completed — Withdrew Consent | 6
Not completed — Investigator Request | 7
Not completed — Other (Unknown) | 3
Period: Long-term Follow-up Period (5 Years)
Arm/Group | Idelalisib
Started | 84 (Participants did not have to complete the TP in order to enter the Long-term Follow-up Period.)
Completed | 20
Not Completed | 64
Not completed — Withdrew Consent | 2
Not completed — Death | 40
Not completed — Lost to Follow-up | 1
Not completed — Other (Unknown) | 21

BASELINE CHARACTERISTICS:
Population: ITT analysis set included enrolled participants who received at least one dose of study drug.
Arm/Group | Idelalisib
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 110
  Race: Black or African American | 2
  Race: Asian | 3
  Race: American Indian or Alaska Native | 1
  Race: Other | 8
  Race: Missing | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 6
  Ethnicity: Not Hispanic or Latino | 117
  Ethnicity: Missing | 2
Region of Enrollment [Count of Participants; unit: Participants]
  France | 10
  United States | 83
  Poland | 8
  Germany | 10
  United Kingdom | 8
  Italy | 6
Karnofsky Performance Status [Count of Participants; unit: Participants] — Karnofsky performance status classified participants according to their functional impairment. Scores ranged from 0-100, the lower the score, the worse the survival for most serious illnesses.
  Participants
    Score = 60 | 2
    Score = 70 | 6
    Score = 80 | 27
    Score = 90 | 44
    Score = 100 | 46
Baseline Disease History [Count of Participants; unit: Participants] — LPL/WM: Lymphoplasmacytic lymphoma/Waldenstrom macroglobulinemia
  Participants
    Folicular lymphoma | 72
    Small lymphocytic lymphoma | 28
    LPL/WM | 10
    Marginal zone lymphoma | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) was assessed based on the International Working Group Revised Response Criteria for Malignant Lymphoma (Cheson, 2007), and was defined as the percentage of participants achieving a complete response (CR) or partial response (PR; or minor response [MR] for participants with WM) as assessed by the study independent review committee (IRC).
  CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
  PR was defined as a ≥ 50% reduction in the sum of the products of the longest perpendicular diameters of all index lesions, with no new lesions.
  For WM only, response was defined as a reduction in immunoglobulin M (IgM) of ≥ 50% decrease for PR, and ≥ 25% decrease for MR; no increase from baseline in the sum of the products of the longest perpendicular diameters of all index lesions, with no new lesions or signs and symptoms of active disease (Owen, 2013)
Time Frame: Start of Treatment to End of Treatment (up to 81 months)
Population: ITT Analysis Set included enrolled participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 125
percentage of participants | 57.6 [48.4 to 66.4]
Statistical Analysis 1: Comparison: Idelalisib; Test type: Superiority; p < 0.0001, Exact binomial test — The null hypothesis is ≤ 20%

2. Secondary Outcome: Duration of Response
Description: Duration of Response (DOR) was defined as the interval from the first documentation of CR or PR (or MR for participants with WM) to the earlier of the first documentation of disease progression as assessed by the study IRC or death from any cause. DOR was analyzed using Kaplan-Meier (KM) estimates.
Time Frame: Start of Treatment to End of Treatment (up to 81 months)
Population: Participants in the ITT Analysis Set who achieved a CR or PR (or MR for participants with WM) were analyzed.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 72
months | 12.5 [6.2 to 28.6]

3. Secondary Outcome: Lymph Node Response Rate
Description: Lymph node response (LNR) was defined as the percentage of participants who achieved a ≥ 50% decrease from baseline in the sum of the product of the perpendicular diameters (SPD) of measurable index lesions as assessed by the study IRC.
Time Frame: Start of Treatment to End of Treatment (up to 81 months)
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 125
percentage of participants | 56.8 [47.6 to 65.6]

4. Secondary Outcome: Time to Response
Description: Time to response (TTR) was defined as the interval from the start of idelalisib treatment to the first documentation of CR or PR (or MR for participants with WM) as assessed by the study IRC.
Time Frame: Start of Treatment to End of Treatment (up to 81 months)
Population: Participants in the ITT Analysis Set who achieved a CR or PR (or MR for participants with WM) were analyzed.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 72
months | 2.0 [1.8 to 4.2]

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the interval from the start of idelalisib treatment to the earlier of the first documentation of disease progression as assessed by the study IRC or death from any cause. PFS was analyzed using KM estimates.
Time Frame: Start of Treatment to End of Treatment (up to 81 months)
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 125
months | 11.1 [8.3 to 14.0]

6. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time interval from the start of idelalisib treatment to death from any cause. OS was analyzed using KM estimates.
Time Frame: Start of Treatment to Last Long-Term Follow-Up Visit (up to maximum of 7 years)
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 125
months | 48.6 [33.9 to 71.7]

7. Secondary Outcome: Change in Health-Related Quality of Life Using the Functional Assessment of Cancer Therapy: Lymphoma Subscale (FACT-LymS)
Description: Change in health-related quality of life events were reported by participants using the Functional Assessment of Cancer Therapy: Lymphoma Subscale (FACT-LymS) assessment tool. Results are presented as the mean (SD) best change from baseline. The best change from baseline was defined as the highest change score (improvement) after baseline.
  The FACT-LymS is on a scale from 0-60, with higher scores associated with a better quality of life. It incorporates values from 15 questions, each rated 0-4, related to study indications.
Time Frame: Baseline to End of Treatment (up to 81 months)
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Idelalisib
Number analyzed (Participants) | 113
units on a scale | 10.3 (17.08)

8. Secondary Outcome: Change in Karnofsky Performance Status
Description: The change in Karnofsky performance status was reported as the best (highest change score) and worst (lowest change score) change from baseline using the Karnofsky performance criteria. The Karnofsky score classified participants according to their functional impairment. Scores are on a scale from 0-100, the lower the score, the worse the survival for most serious illnesses.
Time Frame: Baseline to End of Treatment (up to 81 months)
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Idelalisib
Number analyzed (Participants) | 122
units on a scale
  Best change | 3.0 (8.71)
  Worst change | -10.7 (12.61)

9. Secondary Outcome: Changes in Plasma Concentrations of Disease-Associated Chemokines and Cytokines
Description: Analysis of the cytokine/chemokine was planned to be performed on a subset of samples from this study along with a subset of samples from other studies. Therefore, data for this Outcome Measure are not reported here because the analysis population includes participants who were not enrolled in this study. ClinicalTrials.gov is designed for reporting results from only those participants who were enrolled in the study and described in the Participant Flow and Baseline Characteristics modules.
Time Frame: Enrollment to End of Treatment (up to 81 months)
Reporting Status: Not Posted

10. Secondary Outcome: Safety and Tolerability of Idelalisib Assessed as the Number of Participants Experiencing Adverse Events (AEs) or Abnormalities in Vital Signs, Laboratory Tests, or Electrocardiograms
Description: This composite endpoint measured the safety and tolerability profile of idelalisib. "Clinically meaningful" abnormalities in vital signs and electrocardiograms (ECG) were as determined by the investigator.
Time Frame: Start of Treatment to End of Treatment (up to 81 months) plus 30 days
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 125
Participants
  Any AE | 123
  AE leading to drug discontinuation | 35
  Serious AE | 72
  Vital signs abnormal - clinically meaningful | 0
  ECG abnormal - clinically meaningful | 0
  Grade 3 or 4 hemoglobin | 2
  Grade 3 or 4 neutrophils | 35
  Grade 3 or 4 platelets | 9
  Grade 3 or 4 alanine aminotransferase | 16
  Grade 3 or 4 aspartate aminotransferase | 11

11. Secondary Outcome: Study Drug Exposure
Description: The average idelalisib exposure was summarized.
Time Frame: Start of Treatment to End of Treatment (up to 81 months)
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 125
months | 13.2 (15.08)

12. Secondary Outcome: Idelalisib Plasma Concentration
Time Frame: Predose and at 1.5 hours (± 5 minutes) postdose on Day 29
Population: Pharmacokinetic (PK) Analysis Set included participants in the ITT Analysis Set who had the necessary baseline and on-study measurements.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 125
ng/mL
  Predose: number analyzed (Participants) | 108
  Predose | 471.6 (486.53)
  Postdose: number analyzed (Participants) | 106
  Postdose | 2187.7 (1050.76)

13. Secondary Outcome: PK Parameter: Cmax
Description: Cmax at Days 1 and 29 was analyzed. Cmax is defined as the maximum concentration of drug.
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose on Days 1 and 29
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 8
ng/mL
  Cmax at Day 1 | 2647.5 (1084.99)
  Cmax at Day 29 | 2258.8 (809.61)

14. Secondary Outcome: PK Parameter: Tmax
Description: Tmax at Days 1 and 29 was analyzed. Tmax is defined as the time of Cmax (the maximum concentration of drug).
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose on Days 1 and 29
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Idelalisib
Number analyzed (Participants) | 8
hours
  Tmax at Day 1 | 1.00 [0.99 to 1.04]
  Tmax at Day 29 | 1.00 [0.95 to 2.00]

15. Secondary Outcome: PK Parameter: AUClast
Description: AUClast at Days 1 and 29 was analyzed. AUClast is defined as the concentration of drug from time zero to the last observable concentration
Time Frame: Predose and at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose on Days 1 and 29
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: hours x ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 8
hours x ng/mL
  AUClast at Day 1 | 9094.76 (2960.391)
  AUClast at Day 29 | 9293.39 (3996.826)

ADVERSE EVENTS:
Time Frame: Adverse Events: Start of Treatment to End of Treatment (up to 81 months) plus 30 days; All-Cause Mortality: Baseline to Last Long-Term Follow-Up Visit (up to maximum of 7 years)
Description: ITT Analysis Set included enrolled participants who received at least one dose of study drug.
Arm/Group | Idelalisib
All-Cause Mortality (participants affected / at risk) | 64/125
Serious Adverse Events (participants affected / at risk) | 72/125
Other Adverse Events (participants affected / at risk) | 123/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=125)
Anaemia (Blood and lymphatic system disorders) | 2
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 3
Splenic infarction (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Visual impairment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Acute abdomen (Gastrointestinal disorders) | 1
Autoimmune colitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 11
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Death (General disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 2
Peripheral swelling (General disorders) | 3
Pyrexia (General disorders) | 15
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Autoimmune disorder (Immune system disorders) | 1
Cellulitis (Infections and infestations) | 1
Cytomegalovirus colitis (Infections and infestations) | 2
Device related infection (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 15
Pneumonia cytomegaloviral (Infections and infestations) | 1
Pneumonia necrotising (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pneumonia pseudomonal (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Sepsis syndrome (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Toxoplasmosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Varicella zoster virus infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Hydronephrosis (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Lymphorrhoea (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=125)
Anaemia (Blood and lymphatic system disorders) | 18
Leukopenia (Blood and lymphatic system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 35
Thrombocytopenia (Blood and lymphatic system disorders) | 23
Abdominal pain (Gastrointestinal disorders) | 21
Abdominal pain upper (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 59
Dysphagia (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 38
Stomatitis (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 20
Asthenia (General disorders) | 14
Chills (General disorders) | 11
Fatigue (General disorders) | 40
Mucosal inflammation (General disorders) | 8
Oedema peripheral (General disorders) | 13
Pain (General disorders) | 9
Pyrexia (General disorders) | 34
Bronchitis (Infections and infestations) | 7
Herpes zoster (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 23
Urinary tract infection (Infections and infestations) | 8
Alanine aminotransferase increased (Investigations) | 18
Aspartate aminotransferase increased (Investigations) | 16
Blood creatinine increased (Investigations) | 9
Blood lactate dehydrogenase increased (Investigations) | 7
Weight decreased (Investigations) | 19
Decreased appetite (Metabolism and nutrition disorders) | 23
Dehydration (Metabolism and nutrition disorders) | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 13
Dizziness (Nervous system disorders) | 11
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 17
Insomnia (Psychiatric disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 40
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 9
Night sweats (Skin and subcutaneous tissue disorders) | 18
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 18
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Statistical Analysis Plan (2013-07-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT01282424/SAP_000.pdf
  • Study Protocol: Amendment 10 (Version 9.0) (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT01282424/Prot_001.pdf